CLINICAL TRIAL: NCT07328516
Title: Natural History Study of Early Life Exposures in Agriculture (ELEA)
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002253; 002253-C
Record Dates: First submitted 2026-01-08; First posted 2026-01-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-23

CONDITIONS: Prostate Cancer; Leukemia; Breast Cancer; Melanoma; Colorectal Cancer
Keywords: Agricultural Health Study; Carolina; National Cancer Institute; Iowa; non-agricultural exposures; Children; Adults; ELEA; National Program of Cancer Registries; Environmental
MeSH Terms: conditions — Prostatic Neoplasms; Leukemia; Breast Neoplasms; Melanoma; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Biological and Adopted Children of parents was formerly in the AHS study: This group consists of individuals who are either biological or adopted children of participants from the original Agricultural Health Study, allowing for examination of intergenerational effects and genetic versus environmental influences.
- Male and Women: This group includes all adult participants, both men and women, reflecting a gender-inclusive cohort that allows for analysis of sex-specific health outcomes and differences.
- Participants who can read and understand consent form: This group includes individuals who are able to comprehend and agree to the study's written consent materials, ensuring informed participation and ethical standards are met.
- Participants who spent time on a farm: This criterion ensures all participants had direct exposure to farm environments during their childhood, providing a basis for studying the impact of early agricultural exposures on long-term health.
- Pregnant Women: Pregnant women are specifically included to ensure that the study can assess health outcomes and potential risks associated with pregnancy in individuals with a background of agricultural exposure.

SUMMARY:
Study Description:

ELEA is an observational cohort study that will collect exposure information and biospecimens from the adult children of the Agricultural Health Study (AHS) cohort (https://aghealth.nih.gov/about; Protocol OH93NCN013).

The primary hypothesis is that early life exposures, particularly those found in the agricultural environment, are associated with cancer and other adverse health outcomes in childhood and early adulthood. Eligible individuals will be invited to complete an online questionnaire. After enrollment, study participants may be asked to donate biological and environmental samples. Participants will be followed for cancer and other disease endpoints. Data will be collected from North Carolina and Iowa health registries, disease specific databases, the National Death Index (NDI), North Carolina and Iowa state health registries, publicly available environmental datasets, discarded sample repository, and collection of available samples. Investigators will access data and biospecimens from the AHS protocol OH93NCN01 and link it to the ELEA population.

In an earlier ELEA protocol (16CN095) the NCI SS IRB approved the protocol to perform linkages. That protocol was closed after the transition to the NIH IRB (per a NHSR determination), but the linkage work continued under the ELEA protocols that remained open with Westat and Iowa.

Objectives:

Primary:

To investigate the effect of specific pesticides and other agricultural exposures and risk of cancer in children and adults.

Secondary:

To investigate the effect of non-agricultural exposures and the risk of cancer and other diseases in children and adults.

Exploratory:

Exploratory objectives include, but are not limited to, the examination of genetic and various molecular biomarkers in relation to childhood agricultural exposures.

Endpoints:

Primary:

Incidence of Cancer

Secondary:

Incidence of diseases other than cancer, survival, and various molecular biomarkers.

DETAILED DESCRIPTION:
Study Description:

ELEA is an observational cohort study that will collect exposure information and biospecimens from the adult children of the Agricultural Health Study (AHS) cohort (https://aghealth.nih.gov/about; Protocol OH93NCN013).

The primary hypothesis is that early life exposures, particularly those found in the agricultural environment, are associated with cancer and other adverse health outcomes in childhood and early adulthood. Eligible individuals will be invited to complete an online questionnaire. After enrollment, study participants may be asked to donate biological and environmental samples. Participants will be followed for cancer and other disease endpoints. Data will be collected from North Carolina and Iowa health registries, disease specific databases, the National Death Index (NDI), North Carolina and Iowa state health registries, publicly available environmental datasets, discarded sample repository, and collection of available samples. Investigators will access data and biospecimens from the AHS protocol OH93NCN01 and link it to the ELEA population.

In an earlier ELEA protocol (16CN095) the NCI SS IRB approved the protocol to perform linkages. That protocol was closed after the transition to the NIH IRB (per a NHSR determination), but the linkage work continued under the ELEA protocols that remained open with Westat and Iowa.

Objectives:

Primary:

To investigate the effect of specific pesticides and other agricultural exposures and risk of cancer in children and adults.

Secondary:

To investigate the effect of non-agricultural exposures and the risk of cancer and other diseases in children and adults.

Exploratory:

Exploratory objectives include, but are not limited to, the examination of genetic and various molecular biomarkers in relation to childhood agricultural exposures.

Endpoints:

Primary:

Incidence of Cancer

Secondary:

Incidence of diseases other than cancer, survival, and various molecular biomarkers.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, aged 18 years old and older.
2. Children (biological or adopted) of an AHS participant ( The Main Agricultural Health Study - A Prospective Study of Cancer and Other Diseases among Men and Women in Agriculture (OH93NCN013)).
3. Spent time on a farm as a child.
4. Ability to understand the written consent information sheet and agree to participate.

EXCLUSION CRITERIA:

There are no exclusionary criteria other than inability to meet the eligibility criteria.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from individuals who meet the following eligibility criteria: males and females, including pregnant women, who are 18 years of age or older; biological or adopted children of a participant in "The Main Agricultural Health Study - A Prospective Study of Cancer and Other Diseases among Men and Women in Agriculture (OH93NCN013)"; individuals who spent time on a farm during their childhood; and those who are able to understand the written consent information sheet and agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 64277 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-12-23 (Estimated); Study Completion 2030-12-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of Cancer | Enrollment over 5 years, ongoing follow-up for life or until study end
  To investigate the effect of specific pesticides and other agricultural exposures on the risk of cancer in children and adults. Participants will complete an online questionnaire (45 60 minutes), provide biological samples, and be monitored for cancer development throughout long-term follow-up.

SECONDARY OUTCOMES:
Incidence of diseases other than cancer, survival, and various molecular biomarkers | Enrollment over 5 years; ongoing follow-up for life or until study end
  To assess the effect of non-agricultural exposures on the risk of cancer and other diseases in children and adults. The study will also track survival and collect molecular biomarker data to better understand additional health outcomes beyond cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Beane Freeman, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metayer C, Colt JS, Buffler PA, Reed HD, Selvin S, Crouse V, Ward MH. Exposure to herbicides in house dust and risk of childhood acute lymphoblastic leukemia. J Expo Sci Environ Epidemiol. 2013 Jul;23(4):363-70. doi: 10.1038/jes.2012.115. Epub 2013 Jan 16. PMID 23321862
- [Background] Patel DM, Jones RR, Booth BJ, Olsson AC, Kromhout H, Straif K, Vermeulen R, Tikellis G, Paltiel O, Golding J, Northstone K, Stoltenberg C, Haberg SE, Schuz J, Friesen MC, Ponsonby AL, Lemeshow S, Linet MS, Magnus P, Olsen J, Olsen SF, Dwyer T, Stayner LT, Ward MH; International Childhood Cancer Cohort Consortium. Parental occupational exposure to pesticides, animals and organic dust and risk of childhood leukemia and central nervous system tumors: Findings from the International Childhood Cancer Cohort Consortium (I4C). Int J Cancer. 2020 Feb 15;146(4):943-952. doi: 10.1002/ijc.32388. Epub 2019 May 24. PMID 31054169
- [Background] Flower KB, Hoppin JA, Lynch CF, Blair A, Knott C, Shore DL, Sandler DP. Cancer risk and parental pesticide application in children of Agricultural Health Study participants. Environ Health Perspect. 2004 Apr;112(5):631-5. doi: 10.1289/ehp.6586. PMID 15064173
- [Background] von Mutius E, Radon K. Living on a farm: impact on asthma induction and clinical course. Immunol Allergy Clin North Am. 2008 Aug;28(3):631-47, ix-x. doi: 10.1016/j.iac.2008.03.010. PMID 18572111
- [Background] Carnes MU, Hoppin JA, Metwali N, Wyss AB, Hankinson JL, O'Connell EL, Richards M, Long S, Freeman LE, Sandler DP, Henneberger PK, Barker-Cummings C, Umbach DM, Thorne PS, London SJ. House Dust Endotoxin Levels Are Associated with Adult Asthma in a U.S. Farming Population. Ann Am Thorac Soc. 2017 Mar;14(3):324-331. doi: 10.1513/AnnalsATS.201611-861OC. PMID 27977294
- [Background] Erber E, Lim U, Maskarinec G, Kolonel LN. Common immune-related risk factors and incident non-Hodgkin lymphoma: the multiethnic cohort. Int J Cancer. 2009 Sep 15;125(6):1440-5. doi: 10.1002/ijc.24456. PMID 19444913
- [Background] Linabery AM, Prizment AE, Anderson KE, Cerhan JR, Poynter JN, Ross JA. Allergic diseases and risk of hematopoietic malignancies in a cohort of postmenopausal women: a report from the Iowa Women's Health Study. Cancer Epidemiol Biomarkers Prev. 2014 Sep;23(9):1903-12. doi: 10.1158/1055-9965.EPI-14-0423. Epub 2014 Jun 24. PMID 24962839